CLINICAL TRIAL: NCT00193687
Title: An Open-Label, Flexible-Dose, Long-Term Safety and Efficacy Study of Bifeprunox in the Treatment of Schizpohrenia (Extension of S154.3.001)
Brief Title: Bifeprunox in the Treatment of Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S154.3.002
Record Dates: First submitted 2005-09-11; First posted 2005-09-19 (Estimated); Last update posted 2008-03-24 (Estimated); Status verified 2008-03

CONDITIONS: Schizophrenia
Keywords: open-label study in the treatment of schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — bifeprunox

INTERVENTIONS:
Drug: bifeprunox

SUMMARY:
Study of the long-term efficacy and safety of bifeprunox in the treatment of schizophrenia. Extension to study S154.3.001.

ELIGIBILITY:
Inclusion Criteria:

diagnosis of schizophrenia, understand nature of study, able to be managed in out-patient setting for long-term bifeprunox treatment

Exclusion Criteria:

current primary diagnosis other than schizophrenia, suicide risk, diagnosis or history of substance abuse, uncontrolled hypertension

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 986 (Actual)
Dates: Start 2005-09; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals